CLINICAL TRIAL: NCT02761083
Title: Post-Marketing Clinical Follow-up (PMCF) Study in Ophthalmic Surgery to Evaluate the Safety and Efficacy of Novosyn® Quick Suture Material. A Multicenter Randomized, Active-controlled, Double-blinded, Prospective, Observational Study.
Brief Title: PMCF-study Using Novosyn® Quick Suture Material in Ophthalmic Surgery
Acronym: OPHTHALNOQ
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Comparator was not available in the planned setting
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAG-O-H-1506
Record Dates: First submitted 2016-05-03; First posted 2016-05-04 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Dacryocystorhinostomy; Ectropion; Entropion; Ptosis; Eyelid Tumor Resection; Blepharoplasty
Keywords: Eye surgery; Suture material; Novosyn Quick; Vicryl Rapid
MeSH Terms: conditions — Ectropion; Entropion; Blepharoptosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Novosyn® Quick (Experimental): Eye surgery using suture material
  Interventions: Device: Novosyn® Quick
- Vicryl® Rapid (Active Comparator): Eye surgery using suture material
  Interventions: Device: Vicryl® Rapid

INTERVENTIONS:
Device: Novosyn® Quick — Eye surgery
  Arms: Novosyn® Quick
Device: Vicryl® Rapid — Eye surgery
  Arms: Vicryl® Rapid

SUMMARY:
The aim of this study is to show that the performance of Novosyn® Quick suture material is comparable with standard suture material used in Ophthalmic surgery. In order to show that, various safety and efficacy parameters have been selected. The outcome regarding these parameters will be compared in 2 treatment groups. Active control group will receive Vicryl® Rapide and the treatment group Novosyn® Quick for ophthalmic surgery. It was decided to design this study as a randomized trial, because limited clinical evidence is available in the literature for the active control group (Vicryl® Rapide) which can be used for comparison. Eye operation will be randomly allocated on the left and right side (1:1) to both treatment groups.

Patients undergoing elective, primary ophthalmic surgery (dacryocystorhinostomy, ectropion, entropion, ptosis, eyelid tumor resection, blepharoplasty)

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an elective, primary ophthalmic surgery for dacryocystorhinostomy, ectropion, entropion, ptosis, eyelid tumor resection, and blepharoplasty.
* Age ≥18 years
* Written informed consent

Exclusion Criteria:

* Emergency surgery
* Previous ophthalmic surgery on the same eye
* Known allergy or inflammation reaction to suture material similar to Vicryl® Rapide or Novosyn® Quíck in previous surgery.
* Cicatrisation base alterations
* Concomitant medication, that might affect wound healing (e.g. immunosuppression therapy, anti-diabetic drugs, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2017-03 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Wound infection rate | 3 months
  Wound infection (Surgical site infection, SSI) is defined according to the definition of the US Centres for Disease Control and Prevention (CDC).
Incidence of Wound dehiscence | until 3 months post-operatively
  A dehiscence of the skin which needs surgical treatment with re-closure
Incidence of Tissue reaction (inflammation) | until 3 months after surgery
  A tissue reaction (inflammation) due to the suture material
Incidence of Suture removal due to adverse events | until 3 months post-operatively
Incidence of Re-suturing due to dehiscence | until 3 months post-operatively
Cumulated frequency of adverse events | until 3 months postoperatively
  (edema, allergic reaction, ulceration, bleeding, granuloma, swelling, recurrence, reoperation, dry eyes)
Pain (VAS) | until 3 months postoperatively
Discomfort (VAS) | until 3 months postoperatively
Scar formation (VAS) | until 3 months postoperatively
Patient satisfaction (VAS) | until 3 months postoperatively
Patient satisfaction (EQ-5D-5L) | until 3 months postoperatively
Cosmetic Result (VAS) | until 3 months postoperatively
Handling of the suture | Intraoperative
  Assessment of the handling of the suture material intra-operatively using a questionnaire including different dimensions (knot security, tensile strength, knot run down, tissue drag etc.) with 5 evaluations levels (excellent, very good, good, satisfied, poor).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Can Misses, Ibiza Town, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No